CLINICAL TRIAL: NCT00879658
Title: A Phase II, Double-blind, Randomized, Multi-center, Adaptive Dose-ranging, Placebo-controlled, Parallel-group Study Evaluating Safety, Tolerability and Efficacy on MRI Lesion Parameters and Determining the Dose Response Curve of BAF312 Given Orally Once Daily in Patients With Relapsing-remitting Multiple Sclerosis.
Brief Title: Safety, Tolerability, Efficacy and Optimal Dose Finding Study of BAF312 in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBAF312A2201; 2008-008719-25 (EudraCT Number)
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis (MS); Relapsing-Remitting; Demyelinating Autoimmune Diseases; Disseminated sclerosis; Encephalomyelitis disseminate; Inflammatory disease; Demyelination; Auto-inflammatory disease; Devic's disease; Balo concentric sclerosis; Schilder's diffuse sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Demyelinating Diseases; Neuromyelitis Optica; Diffuse Cerebral Sclerosis of Schilder | interventions — siponimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- BAF312 10mg (period 1) (Experimental)
  Interventions: Drug: BAF312
- BAF312 2 mg (period 1) (Experimental)
  Interventions: Drug: BAF312
- BAF312 0.5 mg (period 1) (Experimental)
  Interventions: Drug: BAF312
- BAF312 dose between 0.1 to 8 mg period 2 (Experimental)
  Interventions: Drug: BAF312
- BAF312 dose between 0.1 - 8 mg period 2 (Experimental)
  Interventions: Drug: BAF312
- Placebo (period 1, 2) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAF312
  Arms: BAF312 0.5 mg (period 1); BAF312 10mg (period 1); BAF312 2 mg (period 1); BAF312 dose between 0.1 - 8 mg period 2; BAF312 dose between 0.1 to 8 mg period 2
Drug: Placebo
  Arms: Placebo (period 1, 2)

SUMMARY:
The purpose of this study was to determine the dose-response curve for the MRI-based efficacy of BAF312 compared with placebo in patients with Relapsing-Remitting Multiple Sclerosis (RRMS), and to characterize its safety and tolerability for the selection of an optimal dose in a later phase III study.

Study Design Rationale An adaptive design was chosen to characterize the dose response curve of BAF312. In a first period of study ("Period 1"), three doses of BAF312 and placebo were tested for MRI efficacy. Based on an interim analysis (IA) after 3 months of treatment, two additional active doses for period 2 wereselected , thus allowing to optimize the overall determination of the dose response curve with 5 data points of active treatment, and placebo. The doses were kept blinded. The use of Modeling and Simulation allowed to establish the full range and dynamics of the dose-response curve in silico, and hence the definition of the optimal dose for later phase III studies.

The choice of placebo as treatment control was essential to obtain information on the specific compared to non-specific effects of active treatment and provides the best way of evaluating the efficacy and of assessing the true safety and tolerability profile of BAF312. Short-term placebo exposure (6 (Period 1) or 3 (Period 2) months, respectively) was unlikely to lead to longer term differences in outcomes [Polman, 2008]. The use of an adaptive design strategy contributed to a significant reduction of placebo exposure, both in terms of the number of patients and duration, as compared to conventional trial models.

Patients having completed the study within the protocol might be eligible for the Extension Phase study where they receive long-term BAF312 treatment (a separate protocol).

ELIGIBILITY:
Key inclusion Criteria:

* Diagnosis of Multiple Sclerosis (MS) as defined by revised McDonald criteria.
* A relapsing-remitting course of disease with at least 1 documented relapse during the previous year, or 2 documented relapses during the previous 2 years, or a positive gadolinium (Gd)-enhanced MRI scan at screening (in case the first MRI scan obtained at screening is negative, a second scan may be obtained 1 month later.)
* An Expanded Disability Status Scale (EDSS) score of 0-5.0 inclusive at randomization.
* Neurologically stable with no evidence of relapse or corticosteroid treatment within 30 days prior to randomization.
* Patients who decline initiation or continuation of treatment with available disease modifying drugs for MS, for whatever reason, after having been informed about their respective benefits and possible adverse events by the investigator.

Key exclusion Criteria:

* A manifestation of another type of MS than RRMS
* History of chronic disease of the immune system other than MS
* Malignancies, diabetes, significant cardiovascular, pulmonary and hepatic diseases and conditions
* Active infections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2009-03-30 (Actual); Primary Completion 2011-05-04 (Actual); Study Completion 2011-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (62):
- United States (16):
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Centennial, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Elk Grove Village, Illinois
  - Novartis Investigative Site, Grand Rapids, Michigan
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Canada (5):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lengerich
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Wiesbaden
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Veszprém
- Italy (4):
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Norway (3):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Drammen
  - Novartis Investigative Site, Oslo
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (4):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Haseki / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mercier F, Bornkamp B, Ohlssen D, Wallstroem E. Characterization of dose-response for count data using a generalized MCP-Mod approach in an adaptive dose-ranging trial. Pharm Stat. 2015 Jul-Aug;14(4):359-67. doi: 10.1002/pst.1693. Epub 2015 Jun 17. PMID 26083135
- [Derived] Selmaj K, Li DK, Hartung HP, Hemmer B, Kappos L, Freedman MS, Stuve O, Rieckmann P, Montalban X, Ziemssen T, Auberson LZ, Pohlmann H, Mercier F, Dahlke F, Wallstrom E. Siponimod for patients with relapsing-remitting multiple sclerosis (BOLD): an adaptive, dose-ranging, randomised, phase 2 study. Lancet Neurol. 2013 Aug;12(8):756-67. doi: 10.1016/S1474-4422(13)70102-9. Epub 2013 Jun 11. PMID 23764350

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in 297 patients at 73 centers in 12 countries.
Pre-assignment Details: One patient was misrandomized and never received study drug. Patient was included in Participant Flow and Baseline Characteristics but not included in actual enrollment count or Full Analysis Set..
Groups:
- BAF312 10mg (Period 1): 10 mg of BAF given orally o.d. for a period of 6 months
- BAF312 2 mg (Period 1): 2 mg of BAF given orally o.d. for a period of 6 months
- BAF312 0.5 mg (Period 1): 0.5 mg of BAF given orally o.d. for a period of 6 months
- Placebo (Period 1): Placebo given orally o.d. for a period of 6 months
- BAF312 1.25 mg (Period 2): 1.25 mg of BAF given orally o.d. for a period of 3 months
- BAF312 0.25 mg (Period 2): 0.25 mg of BAF given orally o.d. for a period of 3 months
- Placebo (Period 2): Placebo given orally o.d. for a period of 3 months
Period: Overall Study
Arm/Group | BAF312 10mg (Period 1) | BAF312 2 mg (Period 1) | BAF312 0.5 mg (Period 1) | Placebo (Period 1) | BAF312 1.25 mg (Period 2) | BAF312 0.25 mg (Period 2) | Placebo (Period 2)
Started | 50 | 49 | 43 | 46 | 42 | 51 | 16
Completed | 35 | 44 | 36 | 42 | 40 | 50 | 16
Not Completed | 15 | 5 | 7 | 4 | 2 | 1 | 0
Not completed — Abnormal laboratory value(s) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Administrative problems | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 3 | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 2 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — misrandomized (never received study med) | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized Set (RAN) consisted of all patients who were assigned a randomization number. The RAN set was used for a summary of patient disposition and demographics and baseline characteristics. One patient was misrandomized and never received study drug. Demographic data was collected and the patient was included in the randomized set.
Groups:
- Placebo (Period 1): Placebo given orally o.d. for a period of 3 months
- Placebo (Period 2): Placebo given orally o.d. for a period of 6 months
- Total: Total of all reporting groups
Arm/Group | BAF312 10mg (Period 1) | BAF312 2 mg (Period 1) | BAF312 0.5 mg (Period 1) | Placebo (Period 1) | BAF312 1.25 mg (Period 2) | BAF312 0.25 mg (Period 2) | Placebo (Period 2) | Total
Number analyzed (Participants) | 50 | 49 | 43 | 46 | 42 | 51 | 16 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Randomized set
  years | 36.4 (8.43) | 37.4 (8.94) | 36.0 (8.79) | 35.2 (8.75) | 35.4 (8.87) | 37.4 (8.39) | 35.9 (8.24) | 36.3 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomized set
  Participants
    Female | 30 | 34 | 30 | 36 | 31 | 42 | 9 | 212
    Male | 20 | 15 | 13 | 10 | 11 | 9 | 7 | 85

OUTCOME MEASURES:

1. Primary Outcome: Dose Responsiveness of BAF312 Based on the Number of Combined Unique Active MRI Lesions (CUAL)
Description: Combined unique active lesions (CUAL) were defined as new gadolinium [Gd]-enhanced lesions on T1-weighted MRI scans or new or enlarging lesions on T2-weighted MRI scans, without double-counting of lesions.
  ED50 is the dose that gives half of the asymptotic maximum change over placebo. ED90 is the dose that gives 90% of the asymptotic maximum change over placebo.
Time Frame: 3 months of treatment
Population: Full analysis set (FAS) consisted of all patients who received at least one dose of study medication and had no protocol deviation with severity code 0 or 8. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Number (95% Confidence Interval); unit: mg
Groups:
- BAF312/Placebo: The dose response relationship among five doses of BAF312 and placebo during 3 months of treatment in patients with RRMS, as measured by the number of combined unique active [MRI] lesions (CUAL).
Arm/Group | BAF312/Placebo
Number analyzed (Participants) | 296
mg
  Dose achieving 50% reduction | 0.51 [0.19 to 1.34]
  ED50 | 0.83 [0.30 to 2.27]
  ED90 | 7.46 [2.72 to 20.47]

2. Secondary Outcome: Number of Confirmed Relapses - Period 1
Description: confirmed relapse: A relapse was to be confirmed by the Independent Evaluating Physician (examining neurologist) performing the EDSS. It was recommended that this occurred within 7 days of the onset of symptoms. A relapse was confirmed when it was accompanied by an increase of at least half a step (0.5) on the EDSS or an increase of 1 point on two different Functional Systems (FS) of the Expanded Disability Status Scale (EDSS) or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
Time Frame: 6 months
Population: Full analysis set in period I
Measure: Number; unit: Confirmed relapses
Groups:
- BAF312 10mg: 10 mg of BAF given orally o.d.
- BAF312 2 mg: 2 mg of BAF given orally o.d.
- BAF312 0.5 mg: 0.5 mg of BAF given orally o.d.
- Placebo: Placebo given orally o.d.
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
Confirmed relapses | 9 | 5 | 13 | 13
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority; p = 0.148, Mixed Models Analysis — Pairwise comparison and p-values refer to ARR on active treatment compared to placebo. An ARR-ratio <1 favors active treatment; Treatment compared to placebo based on negative binomial regression model, adjusted for treatment group and baseline number of relapses in prev 2 yrs; Negative binomial regression model = 0.524, 95% CI 2-sided [0.219 to 1.257]; An ARR-ratio <1 favors active treatment
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Superiority; p = 0.041, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Negative binomial regression model = 0.340, 95% CI 2-sided [0.121 to 0.956]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; Test type: Superiority; p = 0.899, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Negative binomial regression model = 1.051, 95% CI 2-sided [0.486 to 2.273]

3. Secondary Outcome: Proportion of Participants With Relapse-free Patients - Period 1 + 2
Description: To explore the effect of BAF312 on the proportion of relapse-free patients (confirmed relapses only)
Time Frame: 3 month
Population: Full analysis set - Period I and II
Measure: Number; unit: Proportion of participants
Groups:
- BAF312 1.25 mg: 1.25 mg of BAF given orally o.d.
- BAF312 0.25 mg: 0.25 mg of BAF given orally o.d.
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Proportion of participants | 0.87 | 0.93 | 0.93 | 0.79 | 0.86 | 0.88
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Other — Pairwise comparison of treatments to placebo are based on odds ratios estimated from a logistic regression model adjusted for treatment group and using number of relapses in the previous 2 years as a covariate; p = 0.879, Regression, Logistic; Proportions are estimated from the logistic regression model. - An odds ratio of > 1 indicates an increased odds in favor of the active treatment; Logistic regression model = 0.915, 95% CI 2-sided [0.288 to 2.925]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.399, Regression, Logistic — Proportions are estimated from the logistic regression model. - An odds ratio of > 1 indicates an increased odds in favor of the active treatment; Logistic regression model = 1.745, 95% CI 2-sided [0.484 to 7.167]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.454, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Logistic regression model = 1.697, 95% CI 2-sided [0.438 to 8.296]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.223, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Logistic regression model = 0.509, 95% CI 2-sided [0.166 to 1.511]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.668, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Logistic regression model = 0.785, 95% CI 2-sided [0.253 to 2.392]

4. Secondary Outcome: Proportion of Participants With Relapse-free Patients - Period 1 Only
Description: To explore the effect of BAF312 on the proportion of relapse-free patients (confirmed relapses only)
Time Frame: 6 months
Population: Full analysis set - Period I One patient in the placebo group was misrandomized and never received study medication.
Measure: Number; unit: proportion of participants
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
proportion of participants | 0.84 | 0.92 | 0.77 | 0.72
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.178, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Logistic regression model = 1.996, 95% CI 2-sided [0.731 to 5.669]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.014, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Logistic regression model = 4.120, 95% CI 2-sided [1.328 to 14.681]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.642, Regression, Logistic — [p-value comment as in outcome 3, analysis 2]; Logistic regression model = 1.266, 95% CI 2-sided [0.468 to 3.494]

5. Secondary Outcome: Number of New [Gd]-Enhanced T1 Lesions Monthly - Period 1 +2 at Month 3
Description: Results for Month 1 through Month 3 inclusive include patients from both Period 1 and Period 2. New lesions at a specific visit were assessed relative to the previous scheduled visit scan. The number of lesions of each type was available from the central MRI reader. No derivation was performed. Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 3 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesion
Groups:
- Placebo: Placebo-controlled
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Lesion | 0.2 (0.61) | 0.4 (1.00) | 0.2 (0.48) | 0.9 (2.48) | 0.6 (1.16) | 1.4 (3.11)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Pairwise treatment comparison between different BAF312 dose groups and placebo used a two-sided significance level of 5% without adjusting for multiplicity; Test type: Superiority; p < 0.001, Regression, Logistic; new Gd-enhanced T1 lesions was compared between treatment groups using a negative binomial generalized estimating equation regression model; lesion ratio = 0.138, 95% CI 2-sided [0.047 to 0.408]
Statistical Analysis 2: Comparison: BAF312 2 mg; Pairwise treatment comparison between different BAF312 dose group and placebo used a two-sided significance level of 5% without adjusting for multiplicity; Test type: Superiority; p = 0.012, Regression, Logistic — new Gd-enhanced T1 lesions was compared between treatment groups using a negative binomial generalized estimating equation regression model; lesion ratio = 0.307, 95% CI 2-sided [0.123 to 0.771]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.113, 95% CI 2-sided [0.036 to 0.358]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.021, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.375, 95% CI 2-sided [0.163 to 0.860]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.062, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.478, 95% CI 2-sided [0.220 to 1.037]

6. Secondary Outcome: Number of New [Gd]-Enhanced T1 Lesions Monthly - Period 1 Only at 6 Months
Description: Month 4 through Month 6 include patients from Period 1 only. New lesions at a specific visit were assessed relative to the previous scheduled visit scan.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
lesions | 0.3 (0.57) | 0.4 (0.96) | 1.4 (4.17) | 1.8 (3.09)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — Pairwise treatment comparison between different BAF312 dose group and placebo used a two-sided significance level of 5% without adjusting for multiplicity; p < 0.001, Regression, Logistic; new lesions was compared between treatment groups using a negative binomial generalized estimating equation regression model; Lesion ratio = 0.154, 95% CI 2-sided [0.063 to 0.376]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.005, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.228, 95% CI 2-sided [0.081 to 0.641]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.188, 95% CI 2-sided [0.070 to 0.509]

7. Secondary Outcome: Number of All New Gd-enhanced T1 Lesions - Period 1 +2 at Month 3
Description: The results for Month 1 through Month 3 includes patients from both Period 1 and Period 2. New lesions at a specific visit were assessed relative to the previous scheduled visit scan.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 3 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Lesions | 0.5 (0.99) | 0.8 (1.46) | 0.3 (0.68) | 1.5 (3.92) | 1.0 (1.54) | 2.0 (3.78)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.002, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.279, 95% CI 2-sided [0.124 to 0.628]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.019, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.396, 95% CI 2-sided [0.182 to 0.861]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.154, 95% CI 2-sided [0.059 to 0.400]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.035, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.454, 95% CI 2-sided [0.219 to 0.945]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.087, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.555, 96% CI 2-sided [0.283 to 1.090]

8. Secondary Outcome: Number of All Gd-enhanced T1 Lesions - Period 1 Only at 6 Months
Description: The results for Month 4 through Month 6 inclusive includes patients from Period 1 only. New lesions at a specific visit were assessed relative to the previous scheduled visit scan.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
Lesions | 0.3 (0.77) | 0.6 (1.37) | 1.1 (3.78) | 3.0 (5.88)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.095, 95% CI 2-sided [0.033 to 0.273]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.180, 95% CI 2-sided [0.069 to 0.470]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.173, 95% CI 2-sided [0.069 to 0.434]

9. Secondary Outcome: Number of Monthly New/Enlarging T2 Lesions - Period 1 +2 at 3 Months
Description: The results for Month 1 through Month 3 inclusive include patients from both Period 1 and Period 2. New lesions at a specific visit were assessed relative to the previous scheduled visit scan.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 3 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg (Period 1) | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Lesions | 0.4 (0.99) | 0.4 (1.00) | 0.2 (0.64) | 1.0 (3.08) | 0.8 (1.39) | 1.5 (3.17)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.005, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.259, 95% CI 2-sided [0.100 to 0.670]
Statistical Analysis 2: Comparison: BAF312 2 mg (Period 1) vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.005, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.276, 95% CI 2-sided [0.112 to 0.676]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.118, 95% CI 2-sided [0.034 to 0.409]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.485, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.683, 95% CI 2-sided [0.234 to 1.991]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.142, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.591, 95% CI 2-sided [0.292 to 1.193]

10. Secondary Outcome: Number of Monthly New/Enlarging T2 Lesions - Period 1 Only at 6 Months
Description: Month 4 through Month 6 inclusive include patients from Period 1 only. New lesions at a specific visit were assessed relative to the previous scheduled visit scan.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
Lesions | 0.4 (0.91) | 0.4 (1.18) | 0.9 (2.97) | 2.1 (3.66)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.161, 95% CI 2-sided [0.062 to 0.421]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.197, 95% CI 2-sided [0.074 to 0.527]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = 0.139, Regression, Logistic — [p-value comment as in outcome 5, analysis 2]; lesion ratio = 0.416, 95% CI 2-sided [0.130 to 1.331]

11. Secondary Outcome: Number of Patients Without Any New MRI Disease Activity - Period 1 +2
Description: The proportion of patients who were free of new Gd-enhanced T1 lesions, and/or free of new or enlarging T2 lesions, i.e. free of new MRI activity (CUAL).
Time Frame: 3 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Participants | 15 | 18 | 20 | 13 | 20 | 11
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority; p = 0.227, Regression, Logistic — Calculated using weighted logistic regression model adj. for tx group and baseline number of Gd-enhanced T1 lesions. Weight used is equal to 1 if all post-baseline scans up to month 3 are available and (k-x)/k if x scans out of k scans are missing
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Superiority; p = 0.020, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; Test type: Superiority; p = 0.001, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; Test type: Superiority; p = 0.122, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; Test type: Superiority; p = 0.034, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Number of Patients Without Any New MRI Disease Activity - Period 1 Only
Description: as for outcome 11
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
Participants | 12 | 16 | 11 | 6
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority; p = 0.335, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Superiority; p = 0.022, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; Test type: Superiority; p = 0.124, Regression, Logistic — [p-value comment as in outcome 11, analysis 1]

13. Secondary Outcome: Number of Monthly New Gd-enhanced T1 Lesions With High Baseline Disease Activity - Period 1 +2 at 3 Months
Description: In patients with high baseline disease activity, the relative reduction in new Gd-enhanced T1 lesions compared to placebo at Month 3.
  High baseline disease activity is defined as >=2 Gd-enhanced T1 lesions at baseline.
  The number of lesions of each type was available as such from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 3 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51 | 61
Lesions | 0.5 (0.93) | 0.5 (1.09) | 0.1 (0.53) | 1.5 (3.68) | 1.5 (1.57) | 2.7 (4.47)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — Pairwise comparison of treatments are based on a negative binomial GEE regression model accounting for repeated measures on each patient, adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month (the month number of each lesion count measurement) interaction, using the log link; p = 0.006, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.129, 95% CI 2-sided [0.030 to 0.561]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p = 0.005, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.159, 95% CI 2-sided [0.044 to 0.578]
Statistical Analysis 3: Comparison: BAF312 1.25 mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p = 0.005, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.052, 95% CI 2-sided [0.007 to 0.405]
Statistical Analysis 4: Comparison: BAF312 0.5 mg vs Placebo; Pairwise comparison of treatments are based on a negative binomial GEE regression model accounting for repeated measures on each patient, adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month (the month number of each lesion count measurement) interaction, using the log link; Test type: Superiority; p = 0.019, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.271, 95% CI 2-sided [0.091 to 0.807]
Statistical Analysis 5: Comparison: BAF312 0.25 mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p = 0.169, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.504, 95% CI 2-sided [0.190 to 1.337]

14. Secondary Outcome: Number of Monthly New Gd-enhanced T1 Lesions With High Baseline Disease Activity - Period 1 Only at 6 Months
Description: In patients with high baseline disease activity, the relative reduction in new Gd-enhanced T1 lesions compared to placebo at Month 6. High baseline disease activity is defined as >=2 Gd-enhanced T1 lesions at baseline.
  The number of lesions of each type was available from the central MRI reader. No derivation was performed.
  Lesion ratio (and 95% CI) is set between the estimated number of lesions on active treatment compared to placebo. Estimates are computed at Month 3 and Month 6. New lesions at a specific visit were assessed relative to the previous visit. The computation was based upon the mean number of monthly new [Gd]- enhanced lesions. Month 3 and Month 6 results are based on two negative binomial GEE regression models accounting for repeated measures on a patient. Both models were adjusted for baseline number of Gd-enhanced T1 lesions and treatment group x month interaction, using the log link.
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
Lesions | 0.5 (0.69) | 0.6 (1.16) | 1.4 (4.26) | 2.1 (2.42)
Statistical Analysis 1: Comparison: BAF312 10mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p < 0.001, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.214, 95% CI 2-sided [0.091 to 0.499]
Statistical Analysis 2: Comparison: BAF312 2 mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p = 0.018, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.240, 95% CI 2-sided [0.074 to 0.779]
Statistical Analysis 3: Comparison: BAF312 0.5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 13, analysis 1]; p = 0.006, Regression, Logistic — p-value corresponds to the lesion ratio and 95% CI of lesion ratio for active treatment in comparison to placebo; lesion ratio = 0.231, 95% CI 2-sided [0.081 to 0.653]

15. Secondary Outcome: Number of CUAL - Period 1
Description: Combined unique active lesions (CUAL) are defined as new Gd-enhanced T1 lesions or new or enlarging T2 lesions, withput double counting of lesions at any specific point in time.
Time Frame: 6 months
Population: Full analysis set One patient in the placebo group was misrandomized and never received study medication.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 0.5 mg | Placebo
Number analyzed (Participants) | 50 | 49 | 43 | 45
lesions | 0.4 (1.04) | 0.4 (1.26) | 0.9 (3.42) | 2.0 (2.71)

16. Secondary Outcome: Geometric Mean BAF312 Plasma Trough Concentrations
Description: Geometric mean BAF312 plasma concentrations by treatment and by visit
Time Frame: Month 1, Month 3, Month 6
Population: The PK Analysis Set consisted of all patients who received at least one dose of active BAF 312 study medication. Patients were analyzed according to the treatment received.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- BAF312 1.2.5 mg: 1.25 mg of BAF given orally o.d.
Arm/Group | BAF312 10mg | BAF312 2 mg | BAF312 1.2.5 mg | BAF312 0.5 mg | BAF312 0.25 mg
Number analyzed (Participants) | 50 | 49 | 42 | 43 | 51
ng/ml
  Month 1: number analyzed (Participants) | 41 | 43 | 38 | 39 | 46
  Month 1 | 127.9732 (65.53329) | 25.1777 (15.05116) | 14.0450 (6.61030) | 6.9490 (4.97572) | 2.8167 (1.17863)
  Month 3: number analyzed (Participants) | 37 | 44 | 33 | 39 | 39
  Month 3 | 127.4595 (74.96856) | 23.5143 (12.51344) | 11.8270 (6.53977) | 6.1075 (3.89391) | 2.4897 (1.64555)
  Month 6: number analyzed (Participants) | 33 | 40 | 42 | 35 | 51
  Month 6 | 104.0332 (75.60951) | 23.4480 (19.27251) | NA (NA) — Dose was not analyze at month 6. | 5.307 (2.75235) | NA (NA) — Dose was not analyze at month 6.

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 2.5 years.
Groups:
- BAF312 10 mg: 10 mg of BAF given orally o.d.
Arm/Group | BAF312 10 mg | BAF312 2 mg | BAF312 1.25 mg | BAF312 0.5 mg | BAF312 0.25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 1/42 | 0/43 | 0/51 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/50 | 4/49 | 2/42 | 8/43 | 0/51 | 0/61
Other Adverse Events (participants affected / at risk) | 46/50 | 42/49 | 26/42 | 34/43 | 34/51 | 45/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 10 mg (N=50) | BAF312 2 mg (N=49) | BAF312 1.25 mg (N=42) | BAF312 0.5 mg (N=43) | BAF312 0.25 mg (N=51) | Placebo (N=61)
Atrioventricular block second degree (Cardiac disorders) | 1 | 3 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Benign intracranial hypertension (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Schizophreniform disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312 10 mg (N=50) | BAF312 2 mg (N=49) | BAF312 1.25 mg (N=42) | BAF312 0.5 mg (N=43) | BAF312 0.25 mg (N=51) | Placebo (N=61)
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 3 | 0 | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 14 | 3 | 0 | 1 | 2 | 2
Palpitations (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 2 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 6 | 3 | 1 | 1 | 3
Dry eye (Eye disorders) | 1 | 0 | 1 | 2 | 0 | 0
Eye pain (Eye disorders) | 2 | 2 | 0 | 0 | 0 | 2
Visual impairment (Eye disorders) | 0 | 1 | 0 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 8 | 2 | 3 | 2 | 3 | 2
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 2 | 0 | 3
Chills (General disorders) | 3 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 4 | 4 | 1 | 0 | 5
Hyperthermia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0 | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 7 | 1 | 4
Temperature intolerance (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 2 | 4 | 1 | 1 | 2 | 4
Nasopharyngitis (Infections and infestations) | 9 | 6 | 8 | 11 | 7 | 8
Oral herpes (Infections and infestations) | 2 | 1 | 2 | 1 | 1 | 3
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 2 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 3 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 1 | 3 | 0 | 7
Urinary tract infection (Infections and infestations) | 2 | 2 | 3 | 2 | 1 | 2
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 4 | 1 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 4 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 3 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 13 | 5 | 1 | 5 | 0 | 6
Headache (Nervous system disorders) | 23 | 15 | 5 | 8 | 5 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2
Migraine (Nervous system disorders) | 3 | 2 | 0 | 0 | 3 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 4 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1 | 4 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 2 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.